CLINICAL TRIAL: NCT05784961
Title: Impact of tDCS on Cannabis Craving in Patients With Schizophrenia and Cannabis Use Disorder: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study
Brief Title: Impact of tDCS on Cannabis Craving in Schizophrenia
Acronym: tCCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Noomane Bouaziz, MD, Principal Investigator, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10477M-tCCS
Record Dates: First submitted 2021-10-17; First posted 2023-03-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Cannabis Use Disorder
Keywords: cannabis use disorder; schizophrenia; cannabis; craving
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: tDCS versus sham tDCS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial direct current stimulation (active tDCS) (Experimental): The transcranial direct current stimulation (tDCS) with two elecrodes placed over the scalp: the anode over the L DLPFG and the cathode over the left temporo-parietal junction (L TPJ)
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): Sham Comparator: sham transcranial direct current stimulation tDCS device allows sham stimulation. tDCS device sham technology allows optimum placebo stimulation via the same stimulation impresssion than active stimulation.
  Electrode placement is the same than the active arm
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS will be delivered using this electrode montage: anode on the left dosolateral prefrontal cortex (L DLPFC) using F3 EEG landmark and cathode on the left temporoparietal junction (L TPJ) on the middle point between T3 and P3 EEG landmark.
  The stimulation will be delivered at an intensity of 2 milliamps, for 20 minutes, five times a day, with 20 min inter sessions (it will be carried out on 5 consecutive days from Monday to Friday). Each processing day corresponds to a visit of V2, V3, V4, V5 and V6.

SUMMARY:
This study aims to evaluate the tDCS's impact on cannabis craving in patients with schizophrenia and cannabis addiction disorder.

DETAILED DESCRIPTION:
The authors set up this randomized, double-blind multicenter study. 7 centers are participating in this research. After randomisation, the patient will have either the placebo or stimulation sessions, by tDCS, 5 session per day, for 5 days. The authors use the Marijuana Craving Questionnaire (MCQ) scale to determine the variation in cannabis craving and measure the impact of treatment on craving, as primary outcome.

secondary objectives include assessing the effect of tDCS on the general psychopathology of schizophrenia, cannabis and tobacco addiction, and on cognitive tests assessing attention and risk taking This study will be the first known multicenter study assessing tDCS impact on cannabis craving in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) aged 18-65
2. Patients with schizophrenia according to DSM 5 criteria with Comorbid diagnosis of "cannabis use disorder"
3. Stabilized patients: total score = 80 at initial PANSS score and = 3 at the following PANSS points:

   * conceptual disorganization
   * distrust
   * hallucinatory behaviour
   * Unusual content of thought
4. Patients without any other drug or psychotherapeutic treatment for cannabis dependence ("naive" patients)
5. Reported cannabis use greater than three times per week in the past three years
6. Signed consent to participate in research
7. Affiliation to a French social security scheme
8. Patient fluent in the French language

Exclusion Criteria:

1. Presence of any other psychiatric disorder, as per DSM-5 criteria.
2. Pregnancy, possible pregnancy due to lack of contraception, breastfeeding.
3. Currently active suicidal or self-injurious ideation (suicidal or not)
4. Patients with Serious medical codition
5. Other "moderate" to "severe" addictions, according to DSM 5 criteria (excluding tobacco and coffee).
6. Contraindications to tDCS (presence of intracranial metal material, intracranial hypertension, etc.).
7. Subjects already treated by tDCS
8. Patients under legal guardianship (except under curatorship)
9. Patients under safeguard of justice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Marijuana Craving Questionnaire (MCQ) | At baseline (Visit 2) and Day 5 (Visit 6)
  To asses variation in cannabis craving state. The minimum value is 9 and the maximum value is 63.

SECONDARY OUTCOMES:
Change in Score of the PANSS (Positive and Negative Syndrome Scale) to assess the psychopathology of schizophrenia | At baseline (Visit 2) and Day 2, Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  assessment of schizophrenia psychopathology. The minimum value is 7 and the maximum value is 49 for positive scale and negative scale. For general psychopathology, the minimum value is 16 and the maximum value is 112.
Change in Score of SNS (schizophrenia negative symptoms) to assess negative symptoms | At baseline (Visit 2) and , Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  Assessment of schizophrenia negative symptoms. The total score is the sum of the 20 items, ranging from 0 (no negative symptoms) to 40 (severe negative symptoms).
Change in Score of CGI (Clinical Global Impression) to clinical outcome | At baseline (Visit 2) and, Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  CGI scale assess clinical outcome
Change in VAS score (visual analog scale) to assess the craving to cannabis | At baseline (Visit 2) and Day 2 (Visit 3), Day 3 (Visit 4),Day 4 (Visit 5), Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  Cannabis craving status assessment. It is a ruler from 0 to 10 : 0 = absence of craving, 1-3 = low craving, 4-6 = moderate craving, 7-9 = intense craving, 10 = extreme craving.
Change in VAS score (visual analog scale) to assessed the craving to nicotine | At baseline (Visit 2) and Day 2 (Visit 3), Day 3 (Visit 4),Day 4 (Visit 5), Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  Nicotine craving status assessment. It is a ruler from 0 to 10 : 0 = absence of craving, 1-3 = low craving, 4-6 = moderate craving, 7-9 = intense craving, 10 = extreme craving.
Change in BART Analogue Risk Task score | At baseline (Visit 2) and Day 5 (V6)
  BART Analogue Risk assesses risk taking behavior
change in STROOP Test score | At baseline (Visit 2) and Day 5 (V6)
  Stroop test assesses continuous attention and inhibition abilities
Change in Exhaled carbon monoxide concentration score | At baseline (Visit 2) and Day 5 (V6)
  concentration assessment of monoxide de concentration
Urinary cannabis test | between baseline (Visit 2), Day 5 (Visit 6), 5 weeks (Visit 7), 13 weeks (Visit 8)
  assessemnt of cannabis presence in urine
Cannabis and tobacco use assessement | At baseline (Visit 2), Day 5 (V6), 5 weeks (V7) and 13 weeks (V8)
  Assessment of actual use of cannabis and tobacco (numbers of cigarettes, number of joints
Score to Big Five to assessed the personnality dimensions | Baseline (Visit 2)
  The "Big Five" model or the big five personality factors is a tool for personality assessment : extraversion (E), agreeableness (A), conscientiousness (C), neuroticism (N) and openness (O).It is a taxonomic system that measures personality traits. The Bige Five consists of 44 items which are rated on a five-point likert scale from 1 (disagree a lot) to 5 (agree a lot).
Change in MCQ (Marijuana Craving Questionnaire) | At baseline (Visit 2), (Visite 6),(Visit 7) and 13 weeks (Visite 8)
  The minimum value is 9 and the maximum value is 63.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ch Ville Evrard, Neuilly-sur-Marne
  - Youcef Bencherif, Neuilly-sur-Marne

IPD SHARING:
Plan to Share IPD: No